CLINICAL TRIAL: NCT02178774
Title: Using Non-invasive Near-infrared Spectroscopy and Color Doppler to Evaluate the Relationship Between the Perfusion of Uterus and Gastrocnemius Muscles of the Parturients Receiving Cesarean Section
Brief Title: Evaluation the Perfusion of Uterus and Lower Extremities During Cesarean Section With NIRS and Color Doppler
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201401059RIND
Record Dates: First submitted 2014-06-23; First posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Diagnostic and Monitoring Anesthesiology Devices Associated With Adverse Incidents
Keywords: Near-Infrared Spectroscopy (NIRS); spinal anesthesia; cesarean section
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- parturients: tissue oxymetry

SUMMARY:
Hypotension after spinal anesthesia for cesarean section is one of the most common perioperative issue, with an incidence up to 83%.Hypotension is mainly induced by the associated sympathetic blockade, with a drop of peripheral vascular resistance in the lower extremities and an increase in venous capacitance. Hypotension is a distress for both anesthesiologists and obstetricians as it endangers parturient's hemodynamics and compromises the uteroplacental blood flow. In clinical practice, there are several ways to treat hypotension after spinal anesthesia such as preloading with intravenous fluids and administrating ephedrine. Normotensive maternal blood pressure does neither guarantee the well-being of the fetus nor ensure the tissue perfusion of the parturient. Based on the anatomy and physiology basis, we hypothesize that uterine perfusion under spinal anesthesia would correlate with the perfusion of the lower extremities. To measure the perfusion of the lower extremities, we use a relative new tool, the non-invasive transcutaneous near infrared spectroscopy.

DETAILED DESCRIPTION:
This is a prospective observational study. Parturients who are going to receive an elective cesarean section will be enrolled. Before entering the operating rooms, the parturient enrolled receives the Doppler studies. The external iliac artery is identified and color Doppler is activated to locate the uterine artery crossed the external iliac artery. The probe is stabilized to obtain the maximum flow velocity waveform.The pulsatility index of these three waveforms is calculated and recorded as the baseline. Three minutes after the anesthetics are injected, the same procedures of color Doppler are performed again, and the PI after the spinal anesthesia is recorded.

Tissue (cerebral) oximeter (INVOS Cerebral Oximeter Model 5100B; Somanetics, Troy, MI, USA) is used for the NIRS technique. Two adhesive sensor patches are attached to the parturient. One sensor patch is applied over the the biceps brachii of the upper limb while the other adhere to the medial side of the gastrocnemius muscle. After the oximeter shows a stable reading, the baseline data are recorded. The parturient then receive spinal anesthesia in the right lateral decubitus position. The intrathecal injection consists of 0.5% hyperbaric bupivacaine. NIBP is monitored at 2.5 minutes interval for 30 minutes. Tissue oximeter starts recording every minute right after local anesthetics are injected into the intrathecal space for a total of fifteen minutes.

ELIGIBILITY:
Inclusion Criteria:

* Parturients
* elective cesarean section
* ASA class I or class II

Exclusion Criteria:

* Emergent cesarean section
* Skin lesions over the site of local anesthetic injection
* Skin lesions over the sites where NIRS patches are about to be attached
* Patients with history of being allergic to NIRS patches
* Patients with coagulopathy or other contraindications for spinal anesthesia

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Parturients who are going to receive an elective cesarean section in NTUH will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
tissue oxygen saturation | Tissue oximeter starts recording before and every minute right after local anesthetics are injected into the intrathecal space for a total of fifteen minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yuna Shih, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan